CLINICAL TRIAL: NCT06935760
Title: Optimised Treatment for Hypertension Trial - A Feasibility and Pilot Trial of Fire and Forget Versus Usual Care With Intensive Blood Pressure Monitoring for Optimal Hypertension Care
Brief Title: Optimised Treatment for Hypertension Trial
Acronym: OPTIMISE-BP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01743
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Fires

STUDY DESIGN:
Intervention Model Description: Two-arm open-label decentralised pragmatic randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fire and forget (Experimental): Evidence informed empirical prescribing of blood pressure (BP) lowering therapy without serial BP monitoring. Regimen chosen based on the average BP reduction and lowest risk of adverse effects observed in placebo controlled randomised trials. No further blood pressure measurements after baseline until end of study at 12 weeks.
  Interventions: Other: Fire and forget
- Usual care with intensive BP monitoring (Active Comparator): usual care prescribing by general practitioner enhanced with intensive blood pressure monitoring
  Interventions: Other: Usual care with more intensive BP monitoring

INTERVENTIONS:
Other: Fire and forget — Evidence informed prescription of BP lowering drugs based on the average observed blood pressure (BP) reduction and risk of treatment discontinuation due to adverse effects in double-blind placebo-controlled randomised clinical trials. Clinicians will prescribe BP treatment regimen using generic, established BP lowering medications that will be expected to achieve at least 80% of future systolic BP values under 130 mmHg. Treatment will be delivered remotely through telehealth consultation. Participants will be asked to avoid routine BP measurements after treatment is commenced to avoid misleading chance fluctuations in BP before 12 weeks. Adverse events will be monitored remotely, and treatments can be adjusted according to adverse events but not according to BP measurements
  Arms: Fire and forget
Other: Usual care with more intensive BP monitoring — Participants will follow-up with their usual general practitioner, who will treat participants BP according to local practice guidelines. General practitioners will have access to the same BP lowering medications as the "fire and forget" treatment group. Participants will continue to monitor their BP throughout the 12 week period through home BP monitoring with optional 24 hour ambulatory BP monitoring. Participants will maintain a BP diary and present their BP results to their treating physician.
  Other Names: More BP measures
  Arms: Usual care with intensive BP monitoring

SUMMARY:
This randomized trial compares two prescribing strategies to treat high blood pressure. One approach involves remote treatment informed by randomized trial evidence without regular monitoring of blood pressure ("fire and forget"), whilst the other involves usual care treatment with access to frequent blood pressure monitoring. The study will enrol participants with uncontrolled high blood pressure and randomize participants 1:1 to a "fire and forget" treatment group or a "more blood pressure monitoring" group for a total of 12 weeks. "Fire and forget" involves choosing the most appropriate treatment based on the highest quality evidence (randomized trial data), after which participants will stop measuring blood pressures until the end of study. The "more blood pressure monitoring" group will involve treatment as usual but with the access to frequent and high quality blood pressure monitoring.

The goal of this research is to:

1. determine which prescribing approach is more effective at lowering blood pressure after 12 weeks (end of study)
2. assess the safety, feasibility and acceptability of the two treatment approaches.

DETAILED DESCRIPTION:
RATIONALE FOR TRIAL DESIGN:

Current pharmacological treatment of hypertension involves titration of treatment according to serial BP monitoring. However, BP is intrinsically variable and subject to significant measurement and random error that leads to a notoriously poor signal-to-noise ratio. Accordingly, measurement of BPs within 1 to 2 months of starting BP lowering treatment are not associated with true treatment response, adverse effects or cardiovascular risk reduction. Two contrasting solutions include 1) 'fire and forget' by prescribing BP lowering drugs empirically based on the desired average BP response observed from placebo controlled randomised trials without measuring repeat BP or 2) continue usual care with more intensive BP monitoring to try and improve the signal-to-noise ratio.

OBJECTIVES:

The primary aim is to compare the efficacy of remote empirical prescribing of BP lowering drugs informed by randomised trial data without routine BP monitoring ('fire and forget') versus usual care enhanced with intensive BP monitoring ('intensive BP monitoring').

The secondary aims are to determine if, compared to usual care with intensive BP monitoring, remote empirical treatment of high BP is acceptable to patients, is cost-effective and safe.

PARTICIPANT ELIGIBILITY:

Key Inclusion Criteria:

* Adult aged ≥18 years
* High BP defined as home SBP ≥135 or DBP ≥85 mmHg, either untreated or receiving one or two BP lowering drugs
* Among untreated individuals, indicated for pharmacological treatment of high BP according to 2023 NHF Cardiovascular Risk Management Guidelines

Key Exclusion Criteria:

* Currently receiving three or more BP lowering drugs
* Home SBP ≥155 mmHg for untreated participants
* Home SBP ≥150 mmHg for participants on one BP lowering drug
* Home SBP ≥145 mmHg for participants on two BP lowering drugs
* Baseline eGFR <45 ml/min/m2
* Any abnormalities on baseline electrolytes that would prevent initiation of BP lowering therapy
* Participants with any other medical condition or taking any other concomitant medication which in the opinion of the investigator would make the participant unsuitable for the trial

TRIAL INTERVENTION & RANDOMISATION:

All participants who meet the eligibility criteria for the trial will be randomised (1:1) to:

Fire and forget: Remote evidence informed empirical prescribing of BP lowering therapy without serial BP monitoring. Regimen chosen based on the average BP reduction and lowest risk of adverse effects observed in placebo controlled randomised trials Intensive BP monitoring: usual care as per GP prescribing enhanced with intensive BP monitoring

TRIAL OUTCOMES:

Primary: Mean difference in change in home SBP from baseline to 12 weeks

Secondary:

* Efficacy: Proportion achieving home BP control <135/85 mmHg, difference in change in systolic DBP from baseline to 12 weeks
* Safety: Incidence of adverse events leading to treatment withdrawal, adverse events of special interest such as symptoms of hypotension, and SAEs from baseline to 12 weeks.
* Acceptability: interviews of participants
* Self-reported medication adherence
* Cost-effectiveness: Average total cost per patient achieving BP control

ELIGIBILITY:
Inclusion Criteria:

* Written Informed consent
* Adult aged ≥18 years
* English proficiency
* High BP defined as home SBP ≥135 or DBP ≥85 mmHg, either untreated or receiving one or two BP lowering drugs
* Among untreated individuals, indicated for pharmacological treatment of high BP according to 2023 Australian Heart Foundation Cardiovascular Risk Management Guidelines
* Willing to receive BP lowering drug treatment remotely if treatment is indicated
* Willing to check BP with home monitoring for 12 weeks
* Willing to participate in telehealth visit at baseline and 12 weeks
* Willing to undergo blood tests

Exclusion Criteria:

* Currently receiving three or more BP lowering drugs
* Currently receiving an antihypertensive that is not one of the five major antihypertensive drug classes
* Home SBP ≥155 mmHg for untreated participants
* Home SBP ≥150 mmHg for participants on one BP lowering drug
* Home SBP ≥145 mmHg for participants on two BP lowering drugs
* Baseline eGFR <45 ml/min/m2
* Any abnormalities on baseline electrolytes that would prevent initiation of BP lowering therapy
* Participants with any other medical condition or taking any other concomitant medication which in the opinion of the investigator would make the participant unsuitable for the trial.
* Of childbearing age and not using contraception.
* Planned international travel for next 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-28 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean difference in systolic blood pressure from baseline to 12 weeks | 12 weeks
  Mean difference in change in home SBP from baseline to 12 weeks between the two treamtent groups.

SECONDARY OUTCOMES:
Proportion achieving home SBP <130 mmHg (%) at 12 weeks | 12 weeks
  Proportion achieving home SBP <130 mmHg (%) at 12 weeks
Proportion achieving home BP control <135/85mmHg at 12 weeks | 12 weeks
  Proportion achieving home BP control <135/85mmHg at 12 weeks
Mean difference in change in home DBP from baseline to 12 week | 12 weeks
  Mean difference in change in home DBP from baseline to 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Wang, MD PhD, Principal Investigator — The George Institute
Locations (1):
- The George Institute for Global Health, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No